CLINICAL TRIAL: NCT06158867
Title: Assessing the Efficacy and Safety of the AcusMu Microneedle Patch in Treating Periorbital Wrinkles and Skin Diseases
Brief Title: Confirmatory Study: Assessing the Efficacy and Safety of the AcusMu Microneedle Patch in Treating Periorbital Wrinkles
Status: Completed | Type: Observational
Sponsor: AcusMu Medtech Co., Ltd. (Industry)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 112S0069
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Wrinkle
Keywords: Microneedle patch; Anti-wrinkle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FMD WK
  Interventions: Device: FMD WK
- Placebo

INTERVENTIONS:
Device: FMD WK — micro-needle patches containing active anti-wrinkle ingredients
  Groups: FMD WK

SUMMARY:
The core objective of this study is to validate the safe and efficacious application of the AcusMu microneedle patch (FMD WK) to enhance the appearance of periorbital wrinkle

DETAILED DESCRIPTION:
This clinical study is a randomized, double-blind, split-face clinical trial investigating the efficacy of AcusMu (FMD WK) for the treatment of periorbital wrinkles. Participants will attend a study center for a two-week period and undergo a two-week post-treatment follow-up after their final treatment session. Each day, they will apply one of two test products: (A) micro-needle patches containing active anti-wrinkle ingredients and (B) placebo patches beneath their eyes. The patches will be gently pressed onto the skin for 5-10 seconds and left in place for 2-8 hours, continuing this regimen for 14 days. Dermatologists will conduct evaluations at four time points during the study: on day 0, day 7, day 14, and day 28 (±2 days) from the commencement of the experiment. The evaluation process will include the calculation of a Fine Wrinkle Improvement Index specifically designed for assessing under-eye wrinkles to measure improvements. Non-invasive skin testing equipment will be employed to measure skin conditions and capture skin images for objective data analysis (Wrinkle Index). Additionally, self-assessment questionnaires will be administered to gather insights into participants' perceptions of the efficacy of micro-needle patches with active anti-wrinkle ingredients and placebo patches in improving periorbital wrinkles over the two-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 99 (regardless of race or gender).
* Diagnosed with mild or moderate periorbital wrinkles by a dermatologist.

Exclusion Criteria:

* Participants with open wounds or active infections on their skin.
* Individuals involved in other studies that could interfere with this trial.
* Pregnant, breastfeeding, or planning to become pregnant during the trial.
* Those with significant medical conditions such as cancer, liver disease, diabetes, kidney disease, or cardiovascular disorders.
* Individuals who have undergone alternative treatments for periorbital wrinkles in the past six months (e.g., laser therapy, radiofrequency).
* Participants concurrently receiving alternative treatments for periorbital wrinkles.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 to 99, irrespective of race or gender, and diagnosed with mild to moderate periorbital wrinkles by a dermatologist.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 subjects provided informed consent to participate in this study. Participants were assigned two different types of patches to be applied under the eyes (a split-face study), with one type on each arm: one randomly allocated active anti-wrinkle ingredient patch and one placebo patch. The 12 subjects underwent non-invasive skin testing equipment to record periorbital wrinkle conditions and completed self-assessment questionnaires during their study visit.
Units Other Than Participants: Half-face
Groups:
- FMD WK: Participants received the microneedle patch beneath their eyes (randomly assigned to one side of the face). Upon application, the microneedles penetrate the upper layers of the skin and dissolve in the interstitial fluid, releasing the active anti-wrinkle ingredients. Microneedle patches are painless and can be administered without training, requiring only video or image instructions.
  Micro-needle patches containing active anti-wrinkle ingredients: Each microneedle (MN) patch consists of an array of solid, water-soluble, micron-scale needles that encapsulate the active anti-wrinkle ingredients. These patches can be directly applied to the skin.
- Placebo: Participants received the patch beneath their eyes (randomly assigned to one side of the face). Upon application to the skin, the microneedles penetrate into the skin's upper layers and dissolve in the interstitial fluid, releasing the placebo. Microneedle patches are painless and can be administered without training, requiring only video or image instructions.
  Micro-needle patches containing placebo: Each microneedle (MN) patch consists of an array of solid, water-soluble, micron-scale needles that encapsulate the placebo. These patches can be directly applied to the skin.
Period: Overall Study
Arm/Group | FMD WK | Placebo
Started | 12; 12 Half-face | 12; 12 Half-face
Completed | 12; 12 Half-face | 12; 12 Half-face
Not Completed | 0; 0 Half-face | 0; 0 Half-face

BASELINE CHARACTERISTICS:
Groups:
- FMD WK/Placebo (A Split-Face Study): We recruited 12 participants, each receiving a microneedle patch beneath one eye, randomly assigned to one side of the face. Each participant received both types of patches: one containing active anti-wrinkle ingredients and the other a placebo.
  Microneedle patches are painless, require no training for application, and can be used with only video or image instructions. Each patch contains an array of solid, water-soluble, micron-scale needles that penetrate the skin's upper layers, dissolve in interstitial fluid, and release either the active anti-wrinkle ingredients or placebo.
Arm/Group | FMD WK/Placebo (A Split-Face Study)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.75 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Improvement in Periorbital Wrinkles From Baseline
Description: 1. This is a half-face trial involving two weeks of treatment followed by a two-week post-treatment follow-up.
  2. Improvements in periorbital wrinkles will be assessed using the Wrinkle Severity Rating Scale (WSRS), which ranges from 0 (no wrinkles) to 5 (severe wrinkles). A lower score indicates an improvement in wrinkle severity.
  3. Each participant's treated half-face serves as the unit of measure. Any decrease in the WSRS score from baseline is counted as an improvement.
Time Frame: Over the course of study completion, an average duration of 4 weeks was observed.
Measure: Count of Participants; unit: Participants
Arm/Group | FMD WK | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Week 2 | 10 | 2
  Week 4 | 8 | 2

2. Primary Outcome: Number of Participants With Adverse Reactions
Description: Evaluate through skin response sheets: erythema, pain, swelling, etc.
Time Frame: Over the course of study completion, an average duration of 4 weeks was observed.
Measure: Count of Participants; unit: Participants
Arm/Group | FMD WK | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | FMD WK | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT06158867/Prot_SAP_000.pdf